CLINICAL TRIAL: NCT01256619
Title: Evaluation of an Oral Contraceptive Containing 30 mg Ethinyloestradiol and 150 mg Desogestrel on Women's Health
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Dr.abbas noroozi, BASIR center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 132/793
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Women With PMS
Keywords: Marvelon; PMS; serum Lipids
MeSH Terms: interventions — Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- marvelon (Active Comparator)
  Interventions: Drug: Marvelon

INTERVENTIONS:
Drug: Marvelon — The study was a clinical trial without any control group. Sixty one healthy women were included in the study. The participants had been referred to family planning clinics centers under the supervision of Tehran University of Medical Science. weight and blood pressure were measured for all participants at baseline, at the end of cycle 1, at end of cycle 2, at the end of cycle 3 and at the end of cycle 6. Blood pressure was measured on the right arm with the subject seated after 10 minutes of rest

SUMMARY:
The desogestrel (150 mg) in combination with ethinyl estradiol (EE, 30 mg) is known as Marvelon in European countries. Previous studies revealed that the Marvelon is good and safe for women. As a study from Thailand showed that the Marvelon to be effective and acceptable in Thai women. Moreover compared to Caucasian women, the incidences of irregular bleeding and side effects were apparently lower in these Asian women . Although Marvelon was used in many countries but it's efficacy didn't reported among Iranian women.

ELIGIBILITY:
Inclusion Criteria:

being on married, being within 18-40 years old, having normal Body mass index (ranged from 20 to 27 kg/m2), don't use any OCP during 3 months ago, having a normal menstruation cycle for the last three cycles, having at least one of following mental and behavioural symptoms ( Fatigue, mood changes, lack of energy, irritability, aggression, depression, decreased concentration, decreased social relationships, having a greed and increased appetite to eating food), having at least one of following physical symptoms (Breast sensitivity, swelling and flatulence) and women tend to use OCP for six consecutive months.

Exclusion Criteria:

pregnancy, having Anorexia or Bulimia, doing breastfeeding, smoke cigarette, Taking sleeping pills more than 3 days per month, Injection estrogen, progesterone or androgen during the past 3 months, Contraindications for OCP (including: thrombophlebitis - Severe liver disease - cerebrovascular accident and heart disease - unexplained uterine bleeding - lupus - breast cancer - migraines - sickle cell anemia - Epilepsy - gallbladder disease - kidney problems - varicocele and family history thrombosis).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
serum Lipids | baseline-1 month & 2month & 3month &6month after intervention

SECONDARY OUTCOMES:
PMS | baseline-1 month & 2month & 3month &6month after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences-BASIR center, Tehran, Tehran Province, Iran